CLINICAL TRIAL: NCT00915291
Title: Sound Prescribing Study - Assessing the Impact of Pharmaceutical Marketing and Promotional Practices on Physician Prescribing
Brief Title: Evaluating Effectiveness of Educational Intervention to Help Physicians Address Inappropriate Patient Requests for Direct-to-Consumer Advertised Prescription Medications
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: American Medical Association (Other)
Collaborators: Attorney General Consumer & Prescriber Education Grant (Other)
Responsible Party: Audiey Kao, MD, PhD, American Medical Association
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: AMA-ES62
Record Dates: First submitted 2009-06-05; First posted 2009-06-08 (Estimated); Last update posted 2009-06-08 (Estimated); Status verified 2009-06

CONDITIONS: Lumbosacral Muscle Strain
Keywords: medical education; clinical decisionmaking; pharmaceutical marketing

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No

ARMS (2):
- Usual education (No Intervention): Participants randomized into the "no intervention" arm were not exposed to the web-based educational modules
- Web-based educational modules (Experimental): Participants randomized into the intervention arm were exposed to the web-based educational modules
  Interventions: Other: Web-based educational modules

INTERVENTIONS:
Other: Web-based educational modules — Interactive case-based modules that includes video vignettes of clinical interactions between hypothetical patients interacting with physicians
  Arms: Web-based educational modules

SUMMARY:
The purpose of this study is to determine whether physicians can be educated to better handle inappropriate requests from patients for direct-to-consumer advertised prescription medications.

DETAILED DESCRIPTION:
Since changes in FDA regulation direct-to-consumer advertising (DTCA), pharmaceutical companies have expended increasing resources to market their products to the public. This has led to increased awareness of diseases and potential treatments, but it has also created more public demand for medications that may not be appropriate for a patient's clinical presentation. This study aims to provide physicians with the knowledge and skills required to help them address inappropriate DTCA medication requests from patients.

ELIGIBILITY:
Inclusion Criteria:

* Resident physicians in internal medicine or family medicine specialties at participating study sites

Exclusion Criteria:

* Completed less than 10 months of residency

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2007-05; Primary Completion 2008-10 (Actual); Study Completion 2008-10 (Actual)

PRIMARY OUTCOMES:
Decision to prescribe celecoxib

CONTACTS AND LOCATIONS:
Overall Officials: Audiey C Kao, MD, PhD, Principal Investigator — American Medical Association
Locations (4):
- United States (4):
  - Stanford University School of Medicine, Stanford, California
  - Creighton University School of Medicine, Omaha, Nebraska
  - University of Pennsylvania School of Medicine, Philadelphia, Pennsylvania
  - University of Texas at Houston Medical School, Houston, Texas